CLINICAL TRIAL: NCT02255643
Title: The Relationship Between Motor Threshold and Effective Stimulation Threshold During Motor Cortex Stimulation
Brief Title: Motor Threshold and Motor Cortex Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H14-01258
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Neuropathic Pain
Keywords: motor cortex stimulation; chronic neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- -10% of effective PMT (Experimental): Patients are set to a voltage 10% less than their original PMT at start of study, Changes in PMT settings
  Interventions: Device: Change of PMT setting
- former setting (+/- 0% of PMT) (Active Comparator): Patients are set to their original PMT at start of study, Changes in PMT settings
  Interventions: Device: Change of PMT setting
- +10% of effective PMT (Experimental): Patients are set to a voltage 10% more than their original PMT at start of study, Changes in PMT settings
  Interventions: Device: Change of PMT setting

INTERVENTIONS:
Device: Change of PMT setting — The patients current motor threshold is determined and the patient is set to a new PMT (= new treatment arm)

SUMMARY:
Motor cortex stimulation (MCS) is a form of brain stimulation for patients with neuropathic pain not responsive to medication. An electrode is placed on the surface of the brain and connected to a programmable battery in the chest.

The strength of stimulation can be individually adjusted by changing the voltage of stimulation. A too high voltage will produce side effects (e.g. seizures) while a too low voltage will not provide pain control. The aim of this study is to analyze the optimal stimulation parameters in patients already implanted with a motor cortex stimulation who have received good pain relief. The actual voltage may vary widely between patients but the investigators feel that there may be an "ideal" voltage if it is measured as a percentage of motor threshold (PMT). If motor threshold is the stimulation voltage that can evoke a muscle contraction then a PMT = 80% would be a voltage that was eighty percent of that value. Although the actual voltage may be widely different between patients, the percentage needed may be very similar. The investigators therefore plan to measure the effect of different percentages of PMT in patients already being treated with motor cortex stimulation.

Systematic analysis of the findings of this study might help the individual participant and future patients to better programming and less side effects.

DETAILED DESCRIPTION:
Motor cortex stimulation (MCS) is a form of brain stimulation for patients with medically refractory neuropathic pain. The strength of stimulation can be individually adjusted by changing the voltage of stimulation. Too high voltage will produce side effects (e.g. seizures) while too low voltage will not provide pain control. The aim of this study is to analyze the optimal stimulation parameters in patients already implanted with a motor cortex stimulation who have received good pain relief. The actual voltage may vary widely between patients (because of the individual variations in tissue resistance) but the investigators feel that there may be an "ideal" voltage if it is measured as a percentage of motor threshold (PMT).

If motor threshold is the voltage that can evoke a muscle contraction then a PMT = 80% would be a voltage that was eighty percent of that value. Although the actual voltage may be different between patients, the effective PMT may be similar since it represents a more physiologic measure of stimulation.

Systematic analysis of the findings of this study might help the individual participant and future patients by reducing voltage to the lowest effective setting and reducing the chance of seizures.

Motor cortex stimulation is used in the treatment of neuropathic pain since 1991 but still no guidelines for programming exist and programming is therefore mainly bases on trial and error. This is mostly due to many variables influencing the choice of stimulation parameters and significant individual differences in susceptibility to stimulation. Routinely the motor threshold is determined during programming to identify the superior limit of voltage at which twitching is induced. No stimulation above the motor threshold should be performed as this is known to cause seizures. The voltage of simulation that will be effective for an individual is unknown at the beginning of the treatment.

The investigators try to find the lowest effective voltage because that will reduce the risk of stimulation-induced seizures and prolong the life of the pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient more than 18 years of age
* Chronic neuropathic pain effectively treated with motor cortex stimulation
* Stable medication during the trial
* Willing and able to comply with the study protocol and to return per the follow-up visit schedule and able to provide informed consent.

Exclusion Criteria:

* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* Technical malfunction of the MCS device
* History of seizures
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain measured on the Visual Analogue Scale with different PMT Settings | at the End of each trial period, typically 14 days after changes in PMT Settings

SECONDARY OUTCOMES:
Quality of Life assessment with the SF-36 questionnaire | at the end of each trial period, typically at 14 days

OTHER OUTCOMES:
Pain assessment with the McGill pain questionnaire to record impact of pain | at the end of each trial period, typically 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Honey, MD, DPhil, Principal Investigator — UBC
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Treatment of thalamic pain by chronic motor cortex stimulation. Pacing Clin Electrophysiol. 1991 Jan;14(1):131-4. doi: 10.1111/j.1540-8159.1991.tb04058.x. PMID 1705329
- [Background] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Chronic motor cortex stimulation for the treatment of central pain. Acta Neurochir Suppl (Wien). 1991;52:137-9. doi: 10.1007/978-3-7091-9160-6_37. PMID 1792954
- [Background] Peyron R, Garcia-Larrea L, Deiber MP, Cinotti L, Convers P, Sindou M, Mauguiere F, Laurent B. Electrical stimulation of precentral cortical area in the treatment of central pain: electrophysiological and PET study. Pain. 1995 Sep;62(3):275-286. doi: 10.1016/0304-3959(94)00211-V. PMID 8657427
- [Background] Lima MC, Fregni F. Motor cortex stimulation for chronic pain: systematic review and meta-analysis of the literature. Neurology. 2008 Jun 10;70(24):2329-37. doi: 10.1212/01.wnl.0000314649.38527.93. PMID 18541887